CLINICAL TRIAL: NCT05496842
Title: Veränderungen ausgewählter Funktions- Und Teilhabebezogener Merkmale Bei Post-COVID-Patient*Innen in Folge Einer Pneumologischen Phase II Rehabilitation [Changes in Selected Function- and Participation-related Characteristics in Post-COVID Patients Following Pneumological Phase II Rehabilitation]
Brief Title: Changes in Selected Function- and Participation-related Characteristics in Post-COVID Patients Following Pneumological Phase II Rehabilitation
Status: Completed | Type: Observational
Sponsor: Pensionsversicherungsanstalt (Other)
Responsible Party: Sponsor
Other Study IDs: 0009 Post-COVID
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Post-COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rehabilitation patients with post-COVID-19 Syndrome: This group includes rehabilitation patients with and without respiratory muscle training
  Interventions: Behavioral: Multimodal pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Multimodal pulmonary rehabilitation — The rehabilitation is based on the biopsychosocial ICF model of the WHO. Taking into account the physical and psychological condition of the patients, an individual therapy plan is created that is tailored to the needs of the patients.

SUMMARY:
The aim of this project is to provide insight into the relatively new group of post-COVID patients. On the basis of data collected in routine practice, function- and participation-related patient characteristics of post-COVID patients are first described descriptively. Subsequently, the extent to which selected function- and participation-related parameters change following a pneumological phase II rehabilitation in this group of patients is investigated. Furthermore, the extent of these possible changes will be compared between post-COVID patients who received respiratory muscle training and post-COVID patients who did not receive respiratory muscle training. Patients were not randomized but assigned to conditions based on medical criteria (e.g., initial respiratory muscle strength).

The present project provides insight into participation- and function-related characteristics of a relatively new patient population, enables the observation of changes in these following pneumological phase II rehabilitation and provides differentiated insights into the course of health-related parameters for specific subgroups (respiratory muscle training vs. no respiratory muscle training).

ELIGIBILITY:
Inclusion Criteria:

The study participants were regular patients in a rehabilitation centre. The data basis consists of secondary data collected during routine operation.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Regular patients with post-COVID-19 Syndrome in inpatient rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 779 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 3 weeks of inpatient rehabilitation
  The 6-minute walk test is a standardized tool to assess functional exercise capacity operationalized by the walk distance.
European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) | 3 weeks of inpatient rehabilitation
  The EQ-5D-5L is a general instrument for measuring patient-reported outcomes (PROs), which can be used to assess the quality of life of patients on different dimensions (mobility, self-care, usual activities, pain/discomfort) on a 5-level scale (Min. = 0, Max. = 5). Lower values indicate less impairments in the respective dimensions.
  Moreover, the EQ-5D-5L assesses the patient's self-rated health on a 100 point visual analog scale (Min. = 0, Max. = 100). Lower values indicate less positive ratings of health.
Patient Health Questionnaire-4 (PHQ-4) | 3 weeks of inpatient rehabilitation
  The Patient Health Questionnaire-4 (PHQ-4) operationalizes core criteria for anxiety and depression on a 4 point likert scale (Min. = 0, Max = 4). Lower values indicate less impairments.

CONTACTS AND LOCATIONS:
Overall Officials: David Felder, Mag., Study Chair — Pensionsversicherungsanstalt
Locations (1):
- Rehabilitationszentrum Weyer, Weyer, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No